CLINICAL TRIAL: NCT01401803
Title: Brow Lifting With Dysport
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kenneth Beer (Individual)
Collaborators: Medicis Pharmaceutical Corporation (Industry)
Responsible Party: Sponsor-Investigator, Kenneth Beer, Investigator, Beer, Kenneth R., M.D., PA
Organization: Beer, Kenneth R., M.D., PA (Individual)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrowDysport2011
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Brow Ptosis; Lid Ptosis
Keywords: periorbital; glabella; ptosis; eyelid; brow
MeSH Terms: conditions — Blepharoptosis | interventions — abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dysport (Other): Dysport injections into the glabella and orbicularis oculi muscles with dose based on muscle mass.
  Interventions: Drug: Dysport

INTERVENTIONS:
Drug: Dysport — Patients entering will be based on gender and assessment of the glabella region (including the corrugators, procerus, and medial frontalis muscles). Muscle mass will be graded separately for males and females as +, ++, or+++ (light/small, moderate/medium, or heavy/large). Male patients will receive 0.3 mL to 0.4 mL (60, 70, or 80 units) in five equally divided doses of Dysport™ and female patients will receive 0.25 mL to 0.35 mL (50, 60 or 70 units) in equally divided doses of Dysport™ at 5 designated injection sites in the glabellar region. On (Day0) patients will be treated with Dysport™ 10 to 20 units bilaterally to the depressor component of the orbicularis. The dosing for patients will be based on assessment of orbicularis muscle mass. Patients will receive .05 mL to 0.1 mL (10 or 20 units) in two equally divided doses of Dysport™. Muscle mass will not be graded based upon gender for this region.

SUMMARY:
The purpose of this study is to provide data to assess Dysport™ injections as a treatment therapy for brow ptosis. This study will assess the outcome of brow lifting with use of Dysport.

DETAILED DESCRIPTION:
One of the most common reasons that patients present to both dermatologists and plastic surgeons is for brow and lid ptosis. Although some patients that present for these entities require surgery, most will decline to have surgical intervention. Alternative treatments include brow lifting with botulinum toxins.

Brow lifting with botulinum toxins may be performed by injecting the muscles responsible for brow and lid depression. These muscles include: the corrugators, procerus, medical aspect of the frontalis and the depressor component of the orbicularis oculi muscles. By relaxing these muscles, the brow elevators may be able to lift the brow and help both brow and lid ptosis. This trial is unique as it utilizes Dysport to treat an entire anatomic muscle group (the brow depressors) rather than injecting isolated muscles._

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects of any race, 25-75 years of age
* Mild to Moderate brow ptosis (2 or 3 on a 5-point Brow Positioning Grading Scale)
* Subject has signed the IRB-approved Informed Consent Form and the Authorization for Use and Release of Health and Research Study Information (HIPAA) form prior to any study-related procedures being performed
* Subject is able to follow study instructions and likely to complete all required visits, as assessed by the Treating Investigator
* Subject has had a urine pregnancy test evaluated as negative* within 7 days prior to planned study treatment, has used contraception for at least a month prior to planned study treatment, and agrees to use contraception for the duration of the study
* Subjects of childbearing potential must have a negative urine pregnancy test result at Baseline and practice a reliable method of contraception throughout the study:

A female is considered of childbearing potential unless she is:

* postmenopausal for >12 months prior to study drug administration;
* without a uterus and/or both ovaries; or
* surgically sterile (e.g., tubal ligation) for >6 months prior to study drug administration.

The following methods of contraception, if properly used, are generally considered reliable for females of childbearing potential who may participate in the study:

* hormonal contraceptives† (oral, patch, injection, implant);
* male condom with intra-vaginal spermicide or diaphragm or cervical cap with spermicide;
* vaginal contraceptive ring;
* intrauterine device;
* surgical sterilization (bilateral tubal ligation);
* partner vasectomized††; or
* total sexual abstinence*.

  * Hormonal contraceptives must be started at least 90 days prior to study drug administration, and intra-uterine contraceptive device must be placed at least 30 days prior to study drug administration.

    * Vasectomized >3 months or with a 0 sperm count; * Female subjects of childbearing potential who are not sexually active are not required to practice a reliable method of contraception. They may be enrolled at the Investigator's discretion provided that they are counseled to remain sexually inactive for the duration of the study and understand the possible risks involved in getting pregnant during the study.

Exclusion Criteria:

* Previous injection of botulinum toxin of any serotype within 6 months, Previous injection of semi-permanent fillers in the upper face (i.e. glabella, periorbital, temporal areas) within the last 12 months. Previous injection of permanent fillers in the upper face (i.e. glabella, periorbital, temporal areas) are excluded
* Subjects who are pregnant (positive urine pregnancy test), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control
* Subjects planning a facial cosmetic procedure during the study period or with prior cosmetic procedures (i.e., surgery) or visible scars that may affect the evaluation of response
* Facial asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, thick sebaceous skin, or an inability to substantially lessen upper facial rhytids even by physically spreading them apart
* Previous cosmetic surgery to the upper face (e.g., periorbital surgery, brow lift, eyelid or eyebrow surgery, etc.)
* Laser resurfacing, or soft tissue augmentation in the periocular area in the 12months preceding Visit 1
* Medical condition that may increase their risk of exposure to botulinum toxin including diagnosed Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis, or any other disease that might interfere with neuromuscular function
* Current use of aminoglycoside antibiotics, curare-like agents, or agents that might interfere with neuromuscular (skeletal) function
* Profound atrophy/excessive weakness of muscles in target areas of injection
* History of facial nerve palsy
* Any patients with known autoimmune disease or compromised immune systems ie HIV, AIDS or current chemotherapy
* Infection at the injection site or systemic infection (in this case, postpone study entry until one week following recovery)
* Allergy or sensitivity to any component of Dysport™
* Evidence of recent alcohol or drug abuse
* Medical and/or psychiatric problems that is severe enough to interfere with the study results (Investigator opinion)
* History of poor cooperation, non-compliance with medical treatment, or unreliability
* Exposure to an investigational drug study within 30 days of the Baseline Visit

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Correction of brow ptosis with dysport injection | 6 Months
  Subjects will be assessed using 5-point brow positioning grading scale at baseline, day 14, month 1,2,4 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Beer, M.D., Principal Investigator — Kenneth Beer, M.D.,PA
Locations (1):
- Kenneth R. Beer, M.D., PA, West Palm Beach, Florida, United States

REFERENCES:
- [Result] Flynn TC, Carruthers JA, Carruthers JA, Clark RE 2nd. Botulinum A toxin (BOTOX) in the lower eyelid: dose-finding study. Dermatol Surg. 2003 Sep;29(9):943-50; discussion 950-1. doi: 10.1046/j.1524-4725.2003.29257.x. PMID 12930337
- [Result] Carruthers JA, Lowe NJ, Menter MA, Gibson J, Nordquist M, Mordaunt J, Walker P, Eadie N; BOTOX Glabellar Lines I Study Group. A multicenter, double-blind, randomized, placebo-controlled study of the efficacy and safety of botulinum toxin type A in the treatment of glabellar lines. J Am Acad Dermatol. 2002 Jun;46(6):840-9. doi: 10.1067/mjd.2002.121356. PMID 12063480
- [Result] Carruthers A, Carruthers J, Said S. Dose-ranging study of botulinum toxin type A in the treatment of glabellar rhytids in females. Dermatol Surg. 2005 Apr;31(4):414-22; discussion 422. doi: 10.1111/j.1524-4725.2005.31107. PMID 15871316